CLINICAL TRIAL: NCT02875223
Title: A Phase 1, Open-label, Dose Finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CC-90011 in Subjects With Relapsed and/or Refractory Solid Tumors and Non-Hodgkin's Lymphomas
Brief Title: A Safety and Efficacy Study of CC-90011 in Participants With Relapsed and/or Refractory Solid Tumors and Non-Hodgkin's Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90011-ST-001
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma, Non-Hodgkin; Neoplasms
Keywords: Safety; CC-90011; Advanced unresectable solid Tumors; Low intermediate-grade lung neuroendocrine tumors (Typical and Atypical carcinoids); Neuroendocrine prostate cancer (NEPC); R/R Non-Hodgkin's Lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms | interventions — pulrodemstat besilate; Rifampin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CC-90011 and Rifampicin (Experimental)
  Interventions: Drug: CC-90011; Drug: Rifampicin
- CC-90011 and Itraconazole (Experimental)
  Interventions: Drug: CC-90011; Drug: Itraconazole

INTERVENTIONS:
Drug: CC-90011 — Specified dose on specified days
Drug: Rifampicin — Specified dose on specified days
  Arms: CC-90011 and Rifampicin
Drug: Itraconazole — Specified dose on specified days
  Arms: CC-90011 and Itraconazole

SUMMARY:
Study CC-90011-ST-001 is an open-label, Phase 1, dose escalation and expansion, First-In-Human (FIH) clinical study of CC-90011 in subjects with advanced unresectable solid tumors (enriched for grade 2 NENs, grade 2 NETs and NECs) and R/R NHL (MZL, including extranodal MZL [EMZL], splenic MZL [SMZL], nodal MZL [NMZL], and histologic transformation of MZL). The dose escalation part (Part A) of the study will explore escalating oral doses of CC-90011 to estimate the maximum tolerated dose (MTD) of CC-90011. The expansion part (Part B) will further evaluate the safety and efficacy of CC-90011 administered at or below the MTD in 3 selected expansion cohorts of approximately 10-20 evaluable subjects each, in order to further define the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or unresectable solid tumors including those who have progressed on (or not been able to tolerate due to medical comorbidities or unacceptable toxicity) standard anticancer therapy or for whom no other approved conventional therapy exists
* Eastern Cooperative Oncology Group Performance Status of 0 to 1

Exclusion Criteria:

* Prior autologous stem cell transplant ≤ 3 months before first dose or those who have not recovered
* Symptomatic or uncontrolled ulcers (gastric or duodenal), particularly those with a history of and/or risk of perforation and gastrointestinal tract hemorrhages
* Impaired cardiac function or clinically significant cardiac diseases
* Poor bone marrow reserve as assessed by Investigator

Refer to protocol defined exclusion criteria for parts C and D. Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- France (3):
  - Local Institution - 101, Dijon
  - Local Institution - 102, Marseille
  - Local Institution - 100, Villejuif
- Italy (3):
  - Local Institution - 200, Bologna
  - Local Institution - 201, Milan
  - Local Institution - 202, Milan
- Japan (3):
  - Local Institution - 501, Chuo-ku, Tokyo
  - Local Institution - 502, Koto-Ku, Tokyo
  - Local Institution - 500, Kashiwa
- Spain (4):
  - Local Institution - 400, Barcelona
  - Local Institution - 402, Madrid
  - Local Institution - 404, Madrid
  - Local Institution - 401, Santander
- United Kingdom (2):
  - Local Institution - 300, London
  - Local Institution - 301, Newcastle upon Tyne

REFERENCES:
- [Background] Hollebecque A, Salvagni S, Plummer R, Isambert N, Niccoli P, Capdevila J, Curigliano G, Moreno V, Martin-Romano P, Baudin E, Arias M, Mora S, de Alvaro J, Di Martino J, Parra-Palau JL, Sanchez-Perez T, Aronchik I, Filvaroff EH, Lamba M, Nikolova Z, de Bono JS. Phase I Study of Lysine-Specific Demethylase 1 Inhibitor, CC-90011, in Patients with Advanced Solid Tumors and Relapsed/Refractory Non-Hodgkin Lymphoma. Clin Cancer Res. 2021 Jan 15;27(2):438-446. doi: 10.1158/1078-0432.CCR-20-2380. Epub 2020 Oct 12. PMID 33046517
- [Derived] Hollebecque A, Salvagni S, Plummer R, Niccoli P, Capdevila J, Curigliano G, Moreno V, de Braud F, de Villambrosia SG, Martin-Romano P, Baudin E, Arias M, de Alvaro J, Parra-Palau JL, Sanchez-Perez T, Aronchik I, Filvaroff EH, Lamba M, Nikolova Z, de Bono JS. Clinical activity of CC-90011, an oral, potent, and reversible LSD1 inhibitor, in advanced malignancies. Cancer. 2022 Sep 1;128(17):3185-3195. doi: 10.1002/cncr.34366. Epub 2022 Jun 23. PMID 35737639
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not enrolled in Part C and Part D as the study was terminated early.
Groups:
- Part A 1.25 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received CC-90011 capsule orally once per week of different doses.
- Part A 2.5 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 2.5 mg of CC-90011 capsule orally once per week.
- Part A 5 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 5 mg of CC-90011 capsule orally once per week.
- Part A 10 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 10 mg of CC-90011 capsule orally once per week.
- Part A 20 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 20 mg of CC-90011 capsule orally once per week.
- Part A 40 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 40 mg of CC-90011 capsule orally once per week.
- Part A 60 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 60 mg of CC-90011 capsule orally once per week.
- Part A 80 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 80 mg of CC-90011 capsule orally once per week.
- Part A 120 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 120 mg of CC-90011 capsule orally once per week.
- Part B - Lung NETs - 60 mg: Participants with advanced low/intermediate-grade Lung Neuroendocrine tumors (NETs) received 60 mg of CC-90011 capsule orally once per week.
- Part B - NEPC - 60 mg: Participants with neuroendocrine prostate carcinoma (NEPC) received 60 mg of CC-90011 capsule orally once per week.
- Part B - MZL - 60 mg: Participants with relapsed and/or refractory (R/R) non-Hodgkin lymphoma (NHL) (marginal zone lymphoma [MZL], including extranodal marginal zone lymphoma [EMZL], splenic marginal zone lymphoma [SMZL], nodal marginal zone lymphoma [NMZL], and histologic transformation of marginal zone lymphoma (MZL) received 60 mg of CC-90011 capsule orally once per week.
- Part B - Japanese Cohort - 60 mg: Japanese participants with relapsed and/or refractory (R/R) advanced unresectable solid tumors (including grade 2 neuroendocrine neoplasm [NENs]/NETs) and R/R non-Hodgkin lymphoma (NHLs) (including diffuse large B-cell lymphoma [DLBCL] and follicular lymphoma [FL] or MZL) received 60 mg of CC-90011 capsule orally once per week
Period: Overall Study
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg | Part B - Lung NETs - 60 mg | Part B - NEPC - 60 mg | Part B - MZL - 60 mg | Part B - Japanese Cohort - 60 mg
Started | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4 | 14 | 2 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4 | 14 | 2 | 3 | 6
Not completed — Other reasons | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 2 | 3 | 6
Not completed — Death | 4 | 4 | 3 | 4 | 2 | 3 | 5 | 7 | 3 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg | Part B - Lung NETs - 60 mg | Part B - NEPC - 60 mg | Part B - MZL - 60 mg | Part B - Japanese Cohort - 60 mg | Total
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4 | 14 | 2 | 3 | 6 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 3 | 3 | 5 | 2 | 3 | 8 | 2 | 7 | 2 | 1 | 4 | 45
  >=65 years | 3 | 1 | 3 | 1 | 0 | 4 | 3 | 2 | 2 | 7 | 0 | 2 | 2 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 2 | 1 | 3 | 4 | 3 | 7 | 0 | 1 | 2 | 34
  Male | 1 | 2 | 3 | 2 | 3 | 5 | 3 | 6 | 1 | 7 | 2 | 2 | 4 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 6 | 4 | 5 | 5 | 3 | 7 | 3 | 7 | 1 | 0 | 6 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 7 | 1 | 3 | 0 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 5 | 6 | 4 | 5 | 5 | 3 | 7 | 3 | 7 | 1 | 0 | 0 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 7 | 1 | 3 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Part A - Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Dose-limiting toxicities (DLTs) during dose escalation are defined as follows, occurring within the Cycle 1 (28 days) DLT assessment period, unless clearly unrelated to CC-90011: Any Grade 4 non-hematologic toxicity; any non-hematologic toxicity Grade ≥ 3 except Grade 3 diarrhea, nausea, or vomiting of ≤ 3 days duration, Grade 3 rash resolving to Grade ≤ 2 within 7 days without recurrence, and Grade 3 fatigue resolving to Grade ≤ 2 within 7 days without recurrence. Hematological toxicities include febrile neutropenia, Grade 4 neutropenia > 7 days, Grade 4 thrombocytopenia > 7 days, or Grade ≥ 3 thrombocytopenia with significant bleeding. Any AE necessitating dose reduction during Cycle 1, or any other toxicity deemed dose-limiting by the safety committee. The MTD is the highest dose at which less than 33% of the population treated with CC-90011 suffer a DLT in the first cycle and at least 6 evaluable participants have been treated at this dose.
Time Frame: Cycle 1 (Each cycle is of 28 days)
Population: DLT Evaluable Population includes participants in Part A are evaluable for DLT if they received at least 75% of the total planned dose of CC-90011 during Cycle 1.
Measure: Count of Participants; unit: Participants
Groups:
- Part A 1.25 mg: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received 1.25 mg of CC-90011 capsule orally once per week.
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 6 | 6 | 9 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4

2. Secondary Outcome: Part A - Clinical Benefit Rate (CBR) as Per Confirmed Best Overall Response Based on Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (RECIST 1.1)
Description: The Clinical benefit rate (CBR) is defined as percentage of participants with tumor responses (as assessed by the Investigators) of CR, PR and durable SD (SD of ≥ 4 months duration). Complete response (CR) is defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Stable Disease (SD) is concluded when the response does not qualify for CR, PR or Progression. Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From first dose (Day 1) till disease progression or death due to any cause (up to 803 days)
Population: The Treated Population included all participants who enrolled and received at least 1 dose of CC-90011 and prespecified to be reported for Part A only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
percentage of participants | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 52.2] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 60.2] | 20.0 [0.5 to 71.6] | 50.0 [11.8 to 88.2] | 33.3 [4.3 to 77.7] | 30.0 [6.7 to 65.2] | 0.0 [0.0 to 60.2]

3. Secondary Outcome: Part A - Objective Response Rate as Per Confirmed Best Overall Response Based on Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (RECIST 1.1)
Description: The Objective Response Rate (ORR) is defined as the percentage of participants whose best response is CR or PR. Complete response (CR) is defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From first dose (Day 1) untill disease progression or death due to any cause (up to 803 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
percentage of participants | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 60.2]

4. Secondary Outcome: Part A - Duration of Response (DoR) Based on Confirmed Responses
Description: Duration of response is measured from the time when criteria for CR/PR are first met (whichever is first recorded) until the first date at which progressive disease is objectively documented. Complete response (CR) is defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From first dose (Day 1) until disease progression or death due to any cause (up to 803 days)
Population: The Treated Population included all participants who enrolled and received at least 1 dose of CC-90011. Treated Population with Confirmed Best Response of CR or PR. Prespecified to be reported for Part A only.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
months |  |  |  |  |  |  |  | NA [NA to NA] — Not estimated due to inadequate number of events with CR or PR. |

5. Secondary Outcome: Part A - Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from the first dose of CC-90011 to the first occurrence of disease progression or death from any cause based on Kaplan-Meier methodology. Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From first dose (Day 1) until disease progression or death due to any cause (up to 803 days)
Population: The Treated Population included all participants who enrolled and received at least 1 dose of CC-90011. Prespecified to be reported for Part A only.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
days | 96.0 [50.0 to 103.0] | 53.0 [50.0 to 189.0] | 107.0 [22.0 to NA] — Not estimated due to inadequate number of events | 51.5 [22.0 to 106.0] | 588.0 [50.0 to 588.0] | 162.0 [20.0 to NA] — Not estimated due to inadequate number of events | 111.5 [53.0 to NA] — Not estimated due to inadequate number of events | 52.0 [17.0 to 164.0] | 107.0 [61.0 to 238.0]

6. Secondary Outcome: Part A - Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from the first dose of study drug to death due to any cause based on Kaplan-Meier methodology.
Time Frame: From first dose (Day 1) until death due to any cause (up to 803 days)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
days | 315.0 [108.0 to 803.0] | 189.0 [53.0 to 204.0] | 611.0 [78.0 to NA] — Not estimated due to inadequate number of events | 322.5 [114.0 to 593.0] | NA [116.0 to NA] — Not estimated due to inadequate number of events | NA [81.0 to NA] — Not estimated due to inadequate number of events | NA [153.0 to NA] — Not estimated due to inadequate number of events | 139.0 [27.0 to NA] — Not estimated due to inadequate number of events | 238.0 [185.0 to NA] — Not estimated due to inadequate number of events

7. Secondary Outcome: Part A - Maximum Observed Plasma Concentration (Cmax) of CC-90011
Description: Blood samples were collected to assess Cmax. Prespecified to be reported for Part A only.
Time Frame: Day 1 and Day 22 of Cycle 1 (Each cycle consist of 28 days)
Population: The PK Evaluable Population included all participants who enrolled, received at least 1 dose of CC-90011, and had at least 1 measurable concentration of CC-90011. Only participants with data available at the specified timepoints are included in the analysis. Prespecified to be reported for Part A only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
ng/mL
  Cycle 1 Day 1 | 0.4077 (35.18) | 0.8042 (46.38) | 1.520 (39.99) | 2.514 (32.41) | 4.526 (75.80) | 16.28 (40.03) | 23.02 (55.31) | 23.66 (37.60) | 42.03 (45.99)
  Cycle Day 22: number analyzed (Participants) | 4 | 4 | 4 | 3 | 5 | 5 | 5 | 9 | 0
  Cycle Day 22 | 0.4181 (48.30) | 0.7708 (42.21) | 1.651 (45.37) | 3.886 (28.94) | 6.924 (62.53) | 10.85 (29.33) | 20.43 (51.67) | 25.26 (62.11) |

8. Secondary Outcome: Part A - Area Under the Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUCt) of CC-90011
Description: Blood samples were collected to assess AUCt. Prespecified to be reported for Part A only.
Time Frame: Day 1 and Day 22 of Cycle 1 (Each cycle consist of 28 days)
Population: The PK Evaluable Population included all participants who enrolled, received at least 1 dose of CC-90011, and had at least 1 measurable concentration of CC-90011. Only participants with data available at the specified timepoints are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
h*ng/mL
  Cycle 1 Day 1 | 5.806 (55.98) | 24.47 (76.85) | 44.77 (35.77) | 103.07 (42.47) | 179.48 (136.69) | 551.55 (19.29) | 704.82 (60.95) | 849.47 (45.94) | 1736.85 (25.11)
  Cycle Day 22: number analyzed (Participants) | 4 | 4 | 4 | 3 | 5 | 5 | 5 | 9 | 0
  Cycle Day 22 | 11.48 (40.94) | 23.54 (25.12) | 45.30 (46.78) | 125.53 (8.738) | 237.12 (83.11) | 337.92 (30.72) | 625.53 (24.73) | 654.76 (55.42) |

9. Secondary Outcome: Part A - Time to Cmax (Tmax) of CC-90011
Description: Blood samples were collected to assess Tmax. Prespecified to be reported for Part A only.
Time Frame: Day 1 and Day 22 of Cycle 1 (Each cycle consist of 28 days)
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
hours
  Cycle 1 Day 1 | 2.083 [2.050 to 4.000] | 2.017 [2.000 to 4.083] | 4.042 [2.000 to 4.133] | 2.000 [1.917 to 2.000] | 4.183 [4.017 to 6.133] | 4.117 [2.000 to 8.067] | 4.075 [4.000 to 6.000] | 4.042 [3.950 to 6.000] | 3.242 [2.083 to 6.000]
  Cycle Day 22: number analyzed (Participants) | 4 | 4 | 4 | 3 | 5 | 5 | 5 | 9 | 0
  Cycle Day 22 | 2.008 [1.950 to 4.067] | 2.992 [1.983 to 4.017] | 3.917 [1.983 to 4.067] | 4.000 [3.833 to 4.167] | 4.567 [2.000 to 6.000] | 4.067 [4.000 to 6.000] | 3.950 [1.867 to 6.000] | 2.083 [2.000 to 6.000] |

10. Secondary Outcome: Part A - Half-life (t1/2) of CC-90011
Description: Blood samples were collected to assess CL/F. Prespecified to be reported for Part A only.
Time Frame: Day 1 and Day 22 of Cycle 1 (Each cycle consist of 28 days)
Population: as for outcome 8
Measure: Median (Full Range); unit: hour
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
hour
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 5 | 6 | 10 | 4
  Cycle 1 Day 1 | 34.33 [20.93 to 66.63] | 73.07 [41.84 to 83.70] | 79.30 [28.86 to 108.39] | 70.54 [51.66 to 94.99] | 68.35 [48.87 to 105.32] | 59.82 [48.34 to 72.33] | 63.88 [50.57 to 90.40] | 58.52 [46.48 to 79.08] | 67.33 [61.17 to 75.06]
  Cycle Day 22: number analyzed (Participants) | 3 | 4 | 4 | 3 | 5 | 5 | 5 | 9 | 0
  Cycle Day 22 | 77.27 [76.35 to 88.38] | 73.25 [67.30 to 96.45] | 53.62 [25.83 to 82.82] | 72.52 [62.75 to 73.84] | 55.76 [44.35 to 139.08] | 71.88 [41.58 to 92.17] | 61.03 [50.61 to 81.10] | 56.03 [30.47 to 86.98] |

11. Secondary Outcome: Part A - Apparent Clearance (CL/F) of CC-90011
Description: Blood samples were collected to assess CL/F. Prespecified to be reported for Part A only.
Time Frame: Day 1 and Day 22 of Cycle 1 (Each cycle consist of 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hours
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
Litres per hours
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 4 | 5 | 5 | 5 | 10 | 4
  Cycle 1 Day 1 |  | 35.61 (NA) — Not calculated due to 1 participant analyzed. | 95.70 (20.82) | 80.08 (44.68) | 64.69 (79.21) | 63.23 (23.92) | 73.37 (65.85) | 81.99 (50.36) | 57.51 (27.62)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part A- Volume of Distribution (Vz/F) of CC-90011
Description: Blood samples were collected to assess Vz/F. Prespecified to be reported for Part A only.
Time Frame: Day 1 and Day 22 of Cycle 1 (Each cycle consist of 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg
Number analyzed (Participants) | 4 | 5 | 6 | 4 | 5 | 6 | 6 | 10 | 4
Litre
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 4 | 4 | 5 | 5 | 10 | 4
  Cycle 1 Day 1 |  | 3400.66 (NA) — Not calculated due to 1 participant analyzed. | 7814.20 (50.12) | 8076.70 (44.02) | 5734.70 (64.00) | 5506.05 (20.02) | 7245.99 (73.93) | 6984.46 (37.88) | 5598.55 (19.95)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Part B - Clinical Benefit Rate (CBR) as Per Confirmed Best Overall Response Based on Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (RECIST 1.1)
Description: The Clinical Benefit Rate (CBR) is defined as tumor responses (as assessed by the Investigators) of CR, PR and durable SD (SD of ≥ 4 months duration). Complete response (CR) is defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Stable Disease (SD) is concluded when the response does not qualify for CR, PR or Progression. Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From first dose (Day 1) until disease progression or death due to any cause (up to 720 days)
Population: The Treated Population included all participants who enrolled and received at least 1 dose of CC-90011. Prespecified to be reported for Part B only
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B - Lung NETs - 60 mg | Part B - NEPC - 60 mg | Part B - MZL - 60 mg | Part B - Japanese Cohort - 60 mg
Number analyzed (Participants) | 14 | 2 | 3 | 6
percentage of participants | 50.0 [23.0 to 77.0] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 16.7 [0.4 to 64.1]

14. Secondary Outcome: Part B - Objective Response Rate as Per Confirmed Best Overall Response Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (RECIST 1.1)
Description: The Objective Response Rate (ORR) is defined as the percent of participants whose best response is CR or PR. Complete response (CR) is defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From first dose (Day 1) till disease progression or death due to any cause (up to 720 days)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B - Lung NETs - 60 mg | Part B - NEPC - 60 mg | Part B - MZL - 60 mg | Part B - Japanese Cohort - 60 mg
Number analyzed (Participants) | 14 | 2 | 3 | 6
percentage of participants | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 45.9]

15. Secondary Outcome: Part B - Duration of Response (DoR)
Description: as for outcome 4
Time Frame: From first dose (Day 1) until disease progression or death due to any cause (up to 720 days)
Population: The Treated Population included all participants who enrolled and received at least 1 dose of CC-90011. Treated Population with Confirmed Best Response of CR or PR. Prespecified to be reported for Part B only.
Arm/Group | Part B - Lung NETs - 60 mg | Part B - NEPC - 60 mg | Part B - MZL - 60 mg | Part B - Japanese Cohort - 60 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Part B - Progression Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from the first dose of CC-90011 to the first occurrence of disease progression or death from any cause based on Kaplan-Meier methodology Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From first dose (Day 1) until disease progression or death due to any cause (up to 720 days)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part B - Lung NETs - 60 mg | Part B - NEPC - 60 mg | Part B - MZL - 60 mg | Part B - Japanese Cohort - 60 mg
Number analyzed (Participants) | 14 | 2 | 3 | 6
days | 140.5 [51.0 to 176.0] | 38.0 [24.0 to NA] — UL of 95% CI not estimated due to insufficient number of events. | 28.0 [22.0 to NA] — UL of 95% CI not estimated due to insufficient number of events. | 81.5 [26.0 to NA] — UL of 95% CI not estimated due to insufficient number of events.

17. Secondary Outcome: Part B - Overall Survival (OS)
Description: as for outcome 6
Time Frame: From first dose (Day 1) until death due to any cause (up to 720 days)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part B - Lung NETs - 60 mg | Part B - NEPC - 60 mg | Part B - MZL - 60 mg | Part B - Japanese Cohort - 60 mg
Number analyzed (Participants) | 14 | 2 | 3 | 6
days | 720.0 [73.0 to NA] — UL of 95% CI not estimated due to insufficient number of events. | 307.0 [214.0 to NA] — UL of 95% CI not estimated due to insufficient number of events. | NA [147.0 to NA] — Median and UL of 95% CI not estimated due to insufficient number of events. | 180.0 [156.0 to NA] — UL of 95% CI not estimated due to insufficient number of events.

18. Primary Outcome: Part A - Maximum Tolerated Dose (MTDs)
Description: The MTD is the highest dose at which less than 33% of the population treated with CC-90011 suffer a DLT in the first cycle and at least 6 evaluable participants have been treated at this dose. Dose-limiting toxicities (DLTs) during dose escalation are defined as follows, occurring within the Cycle 1 (28 days) DLT assessment period, unless clearly unrelated to CC-90011: Any Grade 4 non-hematologic toxicity; any non-hematologic toxicity Grade ≥ 3 except Grade 3 diarrhea, nausea, or vomiting of ≤ 3 days duration, Grade 3 rash resolving to Grade ≤ 2 within 7 days without recurrence, and Grade 3 fatigue resolving to Grade ≤ 2 within 7 days without recurrence. Hematological toxicities include febrile neutropenia, Grade 4 neutropenia > 7 days, Grade 4 thrombocytopenia > 7 days, or Grade ≥ 3 thrombocytopenia with significant bleeding. Any AE necessitating dose reduction during Cycle 1, or any other toxicity deemed dose-limiting by the safety committee.
Time Frame: Cycle 1 (Each cycle is of 28 days)
Population: as for outcome 1
Measure: Number; unit: milligram
Groups:
- Part A - All DLT Evaluable Participants: Participants with Advanced Solid Tumors and Non-Hodgkin Lymphomas received CC-90011 capsule orally once per week of different doses.
Arm/Group | Part A - All DLT Evaluable Participants
Number analyzed (Participants) | 47
milligram | 60

ADVERSE EVENTS:
Time Frame: All cause mortality was collected in Part A (up to 803 days) and Part B (up to 720 days). Adverse Events (AEs) and Serious AEs were collected from first dose (Day 1) and up to 28 days after last dose for participants in Part A (up to approximately 114 weeks) and Part B (up to approximately 256 weeks).
Description: All cause mortality, serious adverse events and non serious adverse events were collected for all the treated participants. Prespecified to be collected combined for Part B.
Groups:
- Part B 60 mg: Participants with Lung NETs, or NEPC, or MZL received 60 mg of CC-90011 capsule orally once per week.
Arm/Group | Part A 1.25 mg | Part A 2.5 mg | Part A 5 mg | Part A 10 mg | Part A 20 mg | Part A 40 mg | Part A 60 mg | Part A 80 mg | Part A 120 mg | Part B 60 mg
All-Cause Mortality (participants affected / at risk) | 4/4 | 4/5 | 3/6 | 4/4 | 2/5 | 3/6 | 5/6 | 7/10 | 3/4 | 14/25
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/5 | 2/6 | 0/4 | 0/5 | 5/6 | 3/6 | 6/10 | 3/4 | 7/25
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 5/6 | 3/4 | 5/5 | 6/6 | 6/6 | 10/10 | 4/4 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A 1.25 mg (N=4) | Part A 2.5 mg (N=5) | Part A 5 mg (N=6) | Part A 10 mg (N=4) | Part A 20 mg (N=5) | Part A 40 mg (N=6) | Part A 60 mg (N=6) | Part A 80 mg (N=10) | Part A 120 mg (N=4) | Part B 60 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A 1.25 mg (N=4) | Part A 2.5 mg (N=5) | Part A 5 mg (N=6) | Part A 10 mg (N=4) | Part A 20 mg (N=5) | Part A 40 mg (N=6) | Part A 60 mg (N=6) | Part A 80 mg (N=10) | Part A 120 mg (N=4) | Part B 60 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 3 | 0 | 4 | 1 | 2 | 1 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 4 | 4 | 7 | 4 | 16
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 0 | 3 | 1 | 1 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 3 | 2 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 9
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 1 | 4 | 1 | 0 | 1 | 4
Asthenia (General disorders) | 0 | 2 | 1 | 3 | 0 | 1 | 1 | 2 | 1 | 8
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 0 | 3 | 1 | 1 | 3 | 2 | 2
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 2
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 0 | 4
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 4
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypoglossal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT02875223/Prot_SAP_000.pdf